CLINICAL TRIAL: NCT01136356
Title: A Within Subject Comparison of Opioid Withdrawal in Opioid Dependent Individuals
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-08045-9; R01DA008045 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Opioid Abuse; Opioid Dependence
Keywords: opioid pharmacology; buprenorphine; morphine; withdrawal; human research
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine, then Buprenorphine (Experimental): Healthy, out of treatment opioid-dependent residential volunteers (N=7) were randomized to receive morphine (120 mg/day i.m.) administered in four divided doses each day for 9 days (30 mg of morphine four times per day). Participants then underwent an 18-day period of spontaneous opioid withdrawal, during which four double blind i.m. placebo injections were administered daily. After the period of spontaneous withdrawal, participants received buprenorphine (32 mg/day i.m.) administered in four divided doses each day for 9 days (8 mg of buprenorphine four times per day) followed by a second 18-day period of spontaneous withdrawal identical to the withdrawal period described above.
  Interventions: Drug: buprenorphine; Drug: morphine
- Buprenorphine, then Morphine (Experimental): Healthy, out of treatment opioid-dependent residential volunteers (N=7) were randomized to receive buprenorphine (32 mg/day i.m.) administered in four divided doses each day for 9 days (8 mg of buprenorphine four times per day). Participants then underwent an 18-day period of spontaneous withdrawal, during which four double blind i.m. placebo injections were administered daily. After the period of spontaneous withdrawal, participants received morphine (120 mg/day i.m.) administered in four divided doses each day for 9 days (30 mg of morphine four times per day) followed by a second 18-day period of spontaneous withdrawal identical to the withdrawal period described above.
  Interventions: Drug: buprenorphine; Drug: morphine

INTERVENTIONS:
Drug: buprenorphine — parenteral buprenorphine may be administered at multiple times each day
Drug: morphine — parenteral morphine may be administered multiple times each day

SUMMARY:
Buprenorphine is an approved medication for the treatment of opioid dependence. It is typically administered once daily as a sublingual tablet combined with naloxone (i.e., Suboxone). Evidence suggests buprenorphine produces relatively low levels of physical dependence. In addition, some research suggests there is relatively little withdrawal following cessation of chronically administered buprenorphine. This study will examine the spontaneous withdrawal associated with abrupt cessation of buprenorphine compared to morphine in opioid dependent individuals. This study will assess the characteristics and time course of withdrawal using subject-rated and observer-rated measures of opioid withdrawal. Physiologic measures and psychomotor performance will be collected during chronic opioid administration and during placebo administration (i.e., during spontaneous withdrawal). Particular attention will be paid to the differences (if any) in sleep disturbances and withdrawal associated hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Be adults ranging in age from 21-55 years old.
* Be dependent on opioids.
* Be willing to accept or desiring of opioid detoxification.
* He healthy as determined by medical screen, history, and vitals.
* Be without significant psychiatric illness besides drug dependence.
* Be without chronic pain.
* Fluent in English (speaking, writing, and reading).
* Be willing and able to participate.

Exclusion Criteria:

* Previous documented allergy to buprenorphine or morphine.
* Are dependent on other drugs besides opioids and tobacco.
* Have current history of significant use of alcohol or sedative/hypnotics.
* Have evidence of significant medical (e.g., insulin dependent diabetes mellitus) or psychiatric (e.g., schizophrenia) illness.
* Are pregnant (female volunteers will receive a pregnancy test before participation in the study and routinely during the study).
* Have an abnormal or prolongation of the corrected QT interval (QTc) on a baseline electrocardiogram (ECG).
* Are seeking treatment for their substance dependence.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Strain, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Result] Tompkins DA, Smith MT, Mintzer MZ, Campbell CM, Strain EC. A double blind, within subject comparison of spontaneous opioid withdrawal from buprenorphine versus morphine. J Pharmacol Exp Ther. 2014 Feb;348(2):217-26. doi: 10.1124/jpet.113.209478. Epub 2013 Nov 13. PMID 24227768
- See also: A double Blind, within Subjects Comparison of Spontaneous Opioid Withdrawal from Buprenorphine versus Morphine — http://www.ncbi.nlm.nih.gov/pubmed/24227768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study site was an in-patient research-based clinic affiliated with the Johns Hopkins University School of Medicine.
Groups:
- Morphine First, Then Buprenorphine: Participants randomized to receive morphine (120 mg/day i.m.) administered in four divide doses for 9 days. Then underwent an 18-day period of spontaneous withdrawal, during which 4 double blind i.m. placebo injections were administered daily. Then administered using buprenorphine (32 mg/day i.m.) with the same time course
- Buprenorphine First, Then Morphine: Participants randomized to receive buprenorphine (32 mg/day i.m.) administered in four divide doses for 9 days. Then underwent an 18-day period of spontaneous withdrawal, during which 4 double blind i.m. placebo injections were administered daily. Then administered using morphine (120 mg/day i.m.) with the same time course
Period: First Intervention
Arm/Group | Morphine First, Then Buprenorphine | Buprenorphine First, Then Morphine
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: First 18-day Withdrawal
Arm/Group | Morphine First, Then Buprenorphine | Buprenorphine First, Then Morphine
Started | 6 | 6
Completed | 2 | 6
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 0
Period: Second Intervention
Arm/Group | Morphine First, Then Buprenorphine | Buprenorphine First, Then Morphine
Started | 2 | 6
Completed | 2 | 6
Not Completed | 0 | 0
Period: Second 18-day Withdrawal
Arm/Group | Morphine First, Then Buprenorphine | Buprenorphine First, Then Morphine
Started | 2 | 6
Completed | 2 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Within Subjects Design: Participants received both study drugs (buprenorphine and morphine) in a randomized sequence.
Arm/Group | Within Subjects Design
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Peak Opioid Withdrawal Assessed by the Clinical Opiate Withdrawal Scale (COWS)
Description: Clinical Opiate Withdrawal Scale (COWS) is an observer-rated tool for quantifying opioid withdrawal. The scale ranges from 0 to 48: Scores 5 to 12 are mild, 13 to 24 are moderate, 25 to 36 are moderately severe, and over 36 are severe withdrawal. The scores on this repeated measure were analyzed by a two-factor ANOVA for mean peak daily COWS ratings.
Time Frame: Average mean peak opioid withdrawal thirty minutes before and after injection assessed up to 59 days
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Morphine | Buprenorphine
Number analyzed (Participants) | 7 | 7
units on a scale | 12.6 [0 to 48] | 1.3 [0 to 48]

2. Secondary Outcome: Mean Daily Peak Pain Ratings Assessed by the Visual Analog Scale (VAS)
Description: Visual Analog Scale (VAS) measures subjective ratings on pain. The scale on this measurement ranges from 0 being "None" to 100 being "Extremely". The results below reflect the subjective measurements of pain taken from day 0 to day 18 of withdrawal from both morphine and buprenorphine.
Time Frame: Average mean daily peak pain ratings assessed from day 0 to day 18 during the 18 day withdrawal period
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Morphine | Buprenorphine
Number analyzed (Participants) | 7 | 7
units on a scale
  Day 0 Withdrawal | 6.1 [0 to 100] | 2 [0 to 100]
  Day 1 Withdrawal | 29.3 [0 to 100] | 6.3 [0 to 100]
  Day 2 Withdrawal | 51.6 [0 to 100] | 13.3 [0 to 100]
  Day 3 Withdrawal | 33.1 [0 to 100] | 9.4 [0 to 100]
  Day 4 Withdrawal | 29.9 [0 to 100] | 8.6 [0 to 100]
  Day 5 Withdrawal | 20.1 [0 to 100] | 11.4 [0 to 100]
  Day 6 Withdrawal | 20.3 [0 to 100] | 8.6 [0 to 100]
  Day 7 Withdrawal | 11.9 [0 to 100] | 8.6 [0 to 100]
  Day 8 Withdrawal | 6.7 [0 to 100] | 13.6 [0 to 100]
  Day 9 Withdrawal | 17.0 [0 to 100] | 8.6 [0 to 100]
  Day 10 Withdrawal | 13.4 [0 to 100] | 6.3 [0 to 100]
  Day 11 Withdrawal | 4.1 [0 to 100] | 8.3 [0 to 100]
  Day 12 Withdrawal | 11.7 [0 to 100] | 9.1 [0 to 100]
  Day 13 Withdrawal | 7.4 [0 to 100] | 12.7 [0 to 100]
  Day 14 Withdrawal | 6.9 [0 to 100] | 7.9 [0 to 100]
  Day 15 Withdrawal | 15.6 [0 to 100] | 12.9 [0 to 100]
  Day 16 Withdrawal | 3.1 [0 to 100] | 11.6 [0 to 100]
  Day 17 Withdrawal | 7.7 [0 to 100] | 6.7 [0 to 100]
  Day 18 Withdrawal | 5.9 [0 to 100] | 9.4 [0 to 100]

3. Secondary Outcome: Mean Peak Sleep Assessed by Pittsburgh Sleep Quality Index (PSQI)
Description: Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality, total scores range from 0 (better) to 21(worse). The data that has been reported reflects the peak scores on the PSQI during the withdrawal period from both morphine and buprenorphine.
Time Frame: Average mean peak sleep assessed once a week for up to 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Morphine | Buprenorphine
Number analyzed (Participants) | 7 | 7
units on a scale
  Week 2 Withdrawal | 10.3 (1.7) | 5.5 (2)
  Week 3 Withdrawal | 11.3 (2.3) | 6.9 (1.5)

ADVERSE EVENTS:
Groups:
- All Participants: The adverse events were not specified per drug intervention, therefore, the adverse events per interventions is unknown. The data below references the adverse events recorded by licensed nursing personnel during the participants' 59-day protocol in a residential research unit. All participants (N=7) were randomized to receive either buprenorphine (32 mg/day i.m.) or morphine (120 mg/day i.m.) administered in four divided doses each day for 9 days (8 mg of buprenorphine four times per day, or 30 mg of morphine four times per day). Participants then underwent an 18-day period of spontaneous opioid withdrawal, during which four double blind i.m. placebo injections were administered daily. After the period of spontaneous withdrawal, participants received the second opioid administration and spontaneous withdrawal period using the same time course described above.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=12)
Nausea (Gastrointestinal disorders) | 4 (13)
Indigestion (Gastrointestinal disorders) | 3 (14)
Lacrimation Increased (Eye disorders) | 2 (11)
Chills (General disorders) | 2 (10)
Insomnia (Psychiatric disorders) | 4 (12)
Headache (General disorders) | 4 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No